CLINICAL TRIAL: NCT05141877
Title: Impact of Propofol-Based Total Intravenous Anesthesia Versus Anesthesia With Sevoflurane on Long-term Outcomes With Patients Undergoing Elective Craniotomy for Primary Brain Tumors
Brief Title: Influences of Propofol and Sevoflurane Anesthesia in Brain Tumor
Acronym: anesthetics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Tri-Service General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-20210167
Record Dates: First submitted 2021-10-18; First posted 2021-12-02 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Brain Tumor
Keywords: Primary brain tumor; Propofol; Sevoflurane; Survival
MeSH Terms: conditions — Brain Neoplasms | interventions — Propofol; Sevoflurane; Anesthesia, Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol Group (Experimental): The propofol group was both induced and maintained at an effect-site concentration (Ce) of 2.0-4.0 mcg/mL by a target-controlled infusion (TCI) system.
  Interventions: Drug: Propofol
- Sevoflurane group (Experimental): The sevoflurane group was maintained via sevoflurane vaporizer between 1% and 3% (target minimum alveolar concentration of 0.7-1.3).
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — The propofol group was both induced and maintained at an effect-site concentration (Ce) of 2.0-4.0 mcg/mL by a target-controlled infusion (TCI) system.
  Other Names: propofol anesthesia
  Arms: Propofol Group
Drug: Sevoflurane — The sevoflurane group was maintained via sevoflurane vaporizer between 1% and 3% (target minimum alveolar concentration of 0.7-1.3).
  Other Names: inhalation anesthesia
  Arms: Sevoflurane group

SUMMARY:
In the preoperative waiting area, the patients are randomly assigned and divided into two groups according to the allocation sequence table (corresponding to 1:1 randomization) generated by the computer. The propofol group was both induced and maintained at an effect-site concentration (Ce) of 2.0-4.0 mcg/mL by a target-controlled infusion (TCI) system. The sevoflurane group was maintained via sevoflurane vaporizer between 1% and 3% (target minimum alveolar concentration of 0.7-1.3). The following patient data were recorded, the type of anesthesia, sex, age at the time of surgery, preoperative Karnofsky performance status (KPS) score and functional capacity, the postoperative complications within 30 days (according Clavien-Dindo classification), American Society of Anesthesiologists(ASA) physical status scores, tumor size, intraoperative blood loss/transfusion, duration of surgery, duration of anesthesia, total opioid (remifentanil/fentanyl/ propofol) use, postoperative radiation therapy, postoperative chemotherapy, postoperative concurrent chemoradiotherapy, the presence of disease progression, and 6-month, 1-year, and 3-year overall survival and Karnofsky performance status score were recorded.

DETAILED DESCRIPTION:
During the operation, the dose of anesthetic drugs (propofol/ fentanyl /remifentanil and sevoflurane/ cisatracurium/ rocuronium) are adjusted to maintain the mean arterial pressure and heartbeat fluctuations within 20% of the baseline value and Entropy (or BIS) value at 40-60in both groups. The following patient data were recorded, the type of anesthesia, sex, age at the time of surgery, preoperative Karnofsky performance status (KPS) score and functional capacity, the postoperative complications within 30 days (according Clavien-Dindo classification), ASA physical status scores, tumor size, intraoperative blood loss/transfusion, duration of surgery, duration of anesthesia, total opioid (remifentanil/ fentanyl/ propofol) use, postoperative radiation therapy, postoperative chemotherapy, postoperative concurrent chemoradiotherapy, the presence of disease progression, and 6-month, 1-year, and 3-year overall survival and Karnofsky performance status score were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Twenty to eighty-year-old.
2. ASA class I-III.
3. Patients undergoing elective craniotomy for primary brain tumors under general anesthesia.

Exclusion Criteria:

1. Severe mental disorder
2. Poor liver function
3. Pregnant or lactating women
4. Morbidly obese
5. Allergy to any of the drugs used in this study
6. Recurrent tumor or repeat surgery
7. Biopsy cases
8. Incomplete outcome-data
9. Palliative treatment after surgery
10. simultaneous treatment of other malignancies
11. Emergency surgery
12. Presence of other malignant tumors
13. Combined propofol and inhalation anesthesia or other anesthetics, such as ketamine or dexmedetomidine
14. Diagnosed as benign brain tumor
15. cerebellum tumor and pituitary gland tumor.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 6-month
  6-month overall survival
Overall survival | 1-year
  1-year overall survival
Overall survival | 3-year
  3-year overall survival

SECONDARY OUTCOMES:
The presence of disease progression | From the date of surgery until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months"
  cancer recurrence after the surgery
Karnofsky performance status score | Baseline (before the day of surgery)
  to access patients' functional impairment
Postoperative complications within 30 days | The period from the day of surgery until postoperative 30 days
  according to Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Fu Wu, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan